CLINICAL TRIAL: NCT04294355
Title: Artificial Intelligence-assisted Colonoscopy Versus Conventional Colonoscopy for Missed Lesions in the Proximal Colon: A Prospective Multi-center Randomized Study in Asia
Brief Title: Artificial Intelligence-assisted Colonoscopy on Detection of Missed Proximal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Tan Tock Seng Hospital (Other); Institute of Gastroenterology and Hepatology, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: UW 19-713
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Colon Adenoma; Colon Polyp
Keywords: Colonoscopy; Artificial intelligence
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Intervention Model Description: Prospective randomized design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial intelligence-Assisted colonoscopy (Experimental): Tandem colonoscopy of proximal colon assisted with artificial intelligence followed by conventional colonoscopy
  Interventions: Device: Artificial intelligence-Assisted colonoscopy; Procedure: Conventional colonoscopy
- Conventional colonoscopy (Active Comparator): Tandem conventional colonoscopy of proximal colon followed by usual conventional colonoscopy
  Interventions: Procedure: Conventional colonoscopy

INTERVENTIONS:
Device: Artificial intelligence-Assisted colonoscopy — Artificial intelligence-Assisted colonoscopy for detection of colonic polyp
  Arms: Artificial intelligence-Assisted colonoscopy
Procedure: Conventional colonoscopy — Conventional colonoscopy

SUMMARY:
This is a prospective multi-center randomized study is to determine whether the use of artificial intelligence (AI)-assistance could reduce the miss rates of polyps and adenomas in the proximal colon during tandem examination

DETAILED DESCRIPTION:
Centers

1. Queen Mary Hospital, Hong Kong, China (Co-ordinating Center)
2. Tan Tock Seng Hospital, Singapore, Singapore
3. Institute of Gastroenterology and Hepatology, Vietnam Union of Science and Technology Association, Hanoi, Vietnam

Study population

Inclusion:

All adult patients, aged 40 or above, undergoing outpatient colonoscopy in the participating centers will be recruited.

Exclusion:

* history of inflammatory bowel disease
* history of colorectal cancer
* previous bowel resection (apart from appendectomy)
* Peutz-Jeghers syndrome, familial adenomatous polyposis or other polyposis syndromes
* bleeding tendency or severe comorbid illnesses for which polypectomy is considered unsafe.

Post-randomization exclusion:

* Cecum could not be intubated for various reasons
* Boston Bowel Preparation Scale (BBPS) score of the proximal colon is <2

Study design This is a prospective randomized trial comparing the miss rates of proximal colonic lesions by AI assisted colonoscopy or conventional colonoscopy (Fig. 1). The study will be conducted in the Endoscopy Centre of the participating hospitals.

Randomization Eligible patients in each center will be randomly allocated in a 1:1 ratio to undergo tandem colonoscopy of the proximal colon first with AI-assistance and follow by conventional white light colonoscopy (Group 1) or conventional white light colonoscopy without AI assistance follow by conventional colonoscopy (Group 2). Proximal colon refers to colonic segment proximal to the splenic flexure. Randomization will be conducted in blocks of 4 by computer generated random sequences and stratified according to indications of colonoscopy (symptomatic vs screening/surveillance). Patients will be blinded to the group assignment.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients, aged 40 or above, undergoing outpatient colonoscopy in the participating centers will be recruited

Exclusion Criteria:

* history of inflammatory bowel disease
* history of colorectal cancer
* previous bowel resection (apart from appendectomy)
* Peutz-Jeghers syndrome, familial adenomatous polyposis or other polyposis syndromes
* bleeding tendency or severe comorbid illnesses for which polypectomy is considered unsafe.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Proximal adenoma missed rate | One day
  The proportion of patients with missed adenomas detected in the second examination only

SECONDARY OUTCOMES:
Proximal polyp missed rate | One day
  The proportion of patients with missed adenomas detected in the second examination only
Proximal adenoma detection rate | One day
  The proportion of patients with at least one adenoma
Proximal polyp detection | One day
  The proportion of patients with at least one polyp

CONTACTS AND LOCATIONS:
Overall Officials: Ka Luen, Thomas Lui, MBBS, Principal Investigator — Queen Mary Hospital, the University of Hong Kong; Wai Keung Leung, MD, Study Director — Queen Mary Hospital, the University of Hong Kong
Locations (3):
- Queen Mary Hospital, Hong Kong, China
- Tan Tock Seng Hospital, Singapore, Singapore
- Institute of Gastroenterology and Hepatology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lui TKL, Hang DV, Tsao SKK, Hui CKY, Mak LLY, Ko MKL, Cheung KS, Thian MY, Liang R, Tsui VWM, Yeung CK, Dao LV, Leung WK. Computer-assisted detection versus conventional colonoscopy for proximal colonic lesions: a multicenter, randomized, tandem-colonoscopy study. Gastrointest Endosc. 2023 Feb;97(2):325-334.e1. doi: 10.1016/j.gie.2022.09.020. Epub 2022 Oct 5. PMID 36208795